CLINICAL TRIAL: NCT06204432
Title: Efficacy of Adjunctive Sodium Citrate in Smell Retraining for People With Post-Acute Sequelae COVID-19 Olfactory Dysfunction
Brief Title: Sodium Citrate in Smell Retraining for People With Post-COVID-19 Olfactory Dysfunction
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-2829
Record Dates: First submitted 2024-01-10; First posted 2024-01-12 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Long Haul COVID-19; Post-Acute COVID-19 Syndrome; Anosmia; Olfaction Disorders
Keywords: Olfaction disorders; Sodium citrate; COVID-19; Olfactory training
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Anosmia; Olfaction Disorders; COVID-19 | interventions — Sodium Citrate; Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two intervention groups. One will use sodium citrate nasal spray and olfactory training twice a day for 12 weeks. The other will use normal saline nasal spray and olfactory training twice a day for 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, care providers, investigators, and outcome assessors will all be blinded to which study arm a participant is in. Only the compounding pharmacy will have access to the non-blinded group assignments, and they oversee the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal Saline (Placebo Comparator): The Normal Saline arm will use normal saline nasal spray and olfactory training twice a day for 12 weeks.
  Interventions: Drug: Normal Saline; Other: Olfactory Training Kit - "The Olfactory Kit, by AdvancedRx"
- Sodium Citrate (Experimental): The Sodium Citrate arm will use sodium citrate nasal spray and olfactory training twice a day for 12 weeks.
  Interventions: Drug: Sodium Citrate; Other: Olfactory Training Kit - "The Olfactory Kit, by AdvancedRx"

INTERVENTIONS:
Drug: Sodium Citrate — Those randomized to the Sodium Citrate arm will use 1 mL of 2.5% sodium citrate (3.5g/140 mL, pH 7.4, 298 mOsmol/L), 0.5 mL in each nostril, twice a day via an atomizer followed by olfactory training.
  Arms: Sodium Citrate
Drug: Normal Saline — Those randomized to the Normal Saline arm will use 1 mL of normal saline, 0.5 mL in each nostril, twice a day via an atomizer followed by olfactory training.
  Arms: Normal Saline
Other: Olfactory Training Kit - "The Olfactory Kit, by AdvancedRx" — All participants, regardless of study arm they are randomized to, will participate in olfactory training twice a day after use of their nasal spray

SUMMARY:
The goal of this pilot study is to assess the feasibility and impact of using sodium citrate nasal spray as an adjunct to olfactory retraining in participants with long-term post-COVID-19 olfactory dysfunction.

The main questions it aims to answer are:

* Is sodium citrate nasal spray in addition to smell retraining feasible for participants to use in terms of participant need/desire, adherence, and adverse events?
* Does sodium citrate nasal spray in addition to smell retraining further improve smell as compared to normal saline spray and smell retraining?

Participants will:

* Provide consent for enrollment.
* Undergo smell testing via Sniffin' Sticks.
* Use a nasal spray (either sodium citrate or normal saline) followed by olfactory retraining twice a day for 12 weeks.
* Return for follow-up Sniffin' Sticks testing.

Researchers will compare the sodium citrate group and the normal saline group to determine differences in smell improvement.

DETAILED DESCRIPTION:
Background: Loss of sense of smell is a hallmark of COVID-19 infection. While about 80% of post-COVID olfactory dysfunction (OD) will experience some spontaneous recovery within 2 months of initial infection, about 20% will continue to suffer long-term.1 Participants with persistent OD suffer great disability including loss of pleasure with eating leading to weight loss and/or gain and other health risks, including possible dementia. Further, loss of smell may lead to harm, with chief examples of inability to smell gas leaks or food that has gone bad. Currently, use of "smell retraining" is recognized internationally as the most accepted method to treat patients with OD, including post-viral or post-infectious OD.2 Some authors have extrapolated that smell retraining may be of benefit in post-COVID OD, however, data is sparse.3

Increased extracellular calcium has been shown to inhibit the olfaction cascade occurring in the nose by either phosphorylating adenylate cyclase or by interacting and decreasing cyclic nucleotide-gated channels sensitivity to cyclin nucleotides. Several studies have been performed to date using sodium citrate administered as a nasal spray to effectively reduce extracellular calcium resulting in temporary sense of smell benefit in those who have smell loss from a variety of causes, most significantly, post-viral or post-infectious loss (PIOD).

Several studies over the last two decades have examined the effect of sodium citrate on olfactory function in those with OD (mainly post-infectious OD) all of which have shown acute improvement in smell, peaking typically around 1 hour after application.4-7 Most recently, in 2021 Whitcroft et al conducted a controlled clinical trial on 60 PIOD participants. They applied sodium citrate intranasal spray to participants' right nostril for two weeks and olfaction was evaluated by Sniffin' Sticks composite TDI score both before the trial and after 2 weeks of sodium citrate use. They found a significant improvement in TDI score, though not reaching clinical significance. Further, while the proportion of participants reporting parosmia did not change, there was a significant reduction in participants reporting phantosmia.8

The hypothesis is that the administration of sodium citrate to the nasal cavity, providing a temporary improvement in sense of smell, before the performance of smell retraining may augment its effects and yield better recovery in post-COVID-19 OD.

Purpose: The goal of this pilot study is to assess the feasibility and impact of using sodium citrate nasal spray as an adjunct to olfactory retraining in participants with long-term post-COVID-19 olfactory dysfunction.

Participants: Adults (> 18 years) with > 3 months of subjective olfactory loss.

Methods: All participants will undergo initial smell testing with the University of Pennsylvania Smell Identification Test (UPSIT) to confirm smell loss before enrollment.

Following screening and consent, enrollment will involve collecting participant data such as medication allergies, time between COVID-19 infection and smell loss, previous smell loss therapies tried, presence of gustatory dysfunction, and use of paxlovid. Participants; olfaction will then be objectively evaluated using "Sniffin' Sticks," a validated psychophysical tool that allows for more detailed assessment of odor threshold, discrimination, and identification.

Participants will be randomized into two groups and blinded. The Sodium Citrate arm will apply a nasal spray of sodium citrate (0.5 mL per nostril) and then perform olfactory training exercises, twice a day for 12 weeks The Normal Saline arm will apply a spray of normal saline (0.5 mL per nostril) and then perform olfactory training exercises, twice a day for 12 weeks. Olfactory training will involve mindful inhalation of 4 primary odortants (lavender, clove, eucalyptus, and lemon), at least 20 seconds for each.

All materials will be provided by AdvancedRx, who will also perform the randomization to ensure investigators are blind as well. Nasal sprays will be shipped in 1-month quantities and adherence will be checked at the end of each month by assessing the amount of spray left in each bottle. During the 12 weeks, at days 7, 28, and 56, investigators will contact the participants to discuss if any adverse events have occurred.

At the end of the 12 weeks, "Sniffin' Sticks" assessment will be repeated, and results compared within and between the groups. Also, the number of eligible participants encountered, the number enrolled, the number who completed the study, the adherence rate, and the adverse event rates will be assessed within the overarching 1 year study period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male and female, ages greater than or equal to 18 years.
* Patients with persistent olfactory dysfunction originating at the time of a confirmed COVID-19 positive test occurring greater than 3 months ago.
* Ability to use nasal spray and be willing to adhere to the nasal spray and olfactory training regimen

Exclusion Criteria:

* Treatment with another investigational drug or other intervention for olfactory dysfunction within the prior three months.
* Current smoker or inhaled tobacco use within the last three months.
* History of chronic sinusitis or nasal polyps.
* History of olfactory dysfunction following head trauma.
* History of sinus or skull base surgery.
* History of persistent olfactory dysfunction related to any other prior cause other than COVID-19 infection.
* Congenital anosmia.
* Inability to return to UNC Health for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The Number of Eligible Patients | 1 year
  The Number of Eligible Patients Who Meet the Inclusion Criteria
The Proportion of Participants Who Were Enrolled in the Study | 1 year
  The Proportion of Participants Who Were Enrolled in the Study and Completed the First Sniffin' Sticks Test.
The Proportion of Participants Who Complete the Study | 1 year
  The Proportion of Participants Who Complete the 12 Weeks of Smell Retraining With Nasal Spray.
Proportion of Participants Who Report Minor or Severe Adverse Events | 1 year
  The proportion of patients who report minor or severe adverse events during the study.
Adherence Rate Distribution | 1, 4, 8, and 12 weeks
  The distribution of adherence rates (2x / day as instructed, 1x / day, <1x / day).

SECONDARY OUTCOMES:
Change in Sniffin' Sticks Score | Baseline, 12 weeks
  Olfactory testing with Sniffin' Sticks, specifically assessing aspects of olfactory threshold, discrimination, and identification abilities, will be performed after each participant's completion of the intervention.The Sniffin' Sticks assessment is an evaluation of a person's olfactory performance through three subtests, namely the threshold test, identification test, and discrimination test (TDI). The test uses pen-like bodies that contain a fiber stick filled with scents. To perform the test, the cap is removed, and the patient smells the scent on the tip of the pen. The odor threshold test that uses n-butanol and involves a single staircase, the odor discrimination test that presents 16 pairs of odorants and requires triple forced choice, and the odor identification test that presents 16 common odorants and requires multiple forced choice from four verbal items per test odorant. Each test is scored 0 to 16, with 16 representing good olfaction and 0 representing poor olfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Brent A. Senior, MD, FACS, FARS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bacon DR, Onuorah P, Murr A, Wiesen CA, Oakes J, Thorp BD, Zanation AM, Ebert CS Jr, Wohl D, Senior BA, Kimple AJ. COVID-19 related olfactory dysfunction prevalence and natural history in ambulatory patients. Rhinol Online. 2021;4(4):131-139. doi: 10.4193/rhinol/21.034. Epub 2021 Aug 13. PMID 34485883
- [Background] Kattar N, Do TM, Unis GD, Migneron MR, Thomas AJ, McCoul ED. Olfactory Training for Postviral Olfactory Dysfunction: Systematic Review and Meta-analysis. Otolaryngol Head Neck Surg. 2021 Feb;164(2):244-254. doi: 10.1177/0194599820943550. Epub 2020 Jul 14. PMID 32660334
- [Background] Wu TJ, Yu AC, Lee JT. Management of post-COVID-19 olfactory dysfunction. Curr Treat Options Allergy. 2022;9(1):1-18. doi: 10.1007/s40521-021-00297-9. Epub 2022 Jan 4. PMID 35004126
- [Background] Panagiotopoulos G, Naxakis S, Papavasiliou A, Filipakis K, Papatheodorou G, Goumas P. Decreasing nasal mucus Ca++ improves hyposmia. Rhinology. 2005 Jun;43(2):130-4. PMID 16008069
- [Background] Whitcroft KL, Merkonidis C, Cuevas M, Haehner A, Philpott C, Hummel T. Intranasal sodium citrate solution improves olfaction in post-viral hyposmia. Rhinology. 2016 Dec 1;54(4):368-374. doi: 10.4193/Rhino16.054. PMID 27316224
- [Background] Whitcroft KL, Ezzat M, Cuevas M, Andrews P, Hummel T. The effect of intranasal sodium citrate on olfaction in post-infectious loss: results from a prospective, placebo-controlled trial in 49 patients. Clin Otolaryngol. 2017 Jun;42(3):557-563. doi: 10.1111/coa.12789. Epub 2016 Dec 7. PMID 27860366
- [Background] Philpott CM, Erskine SE, Clark A, Leeper A, Salam M, Sharma R, Murty GE, Hummel T. A randomised controlled trial of sodium citrate spray for non-conductive olfactory disorders. Clin Otolaryngol. 2017 Dec;42(6):1295-1302. doi: 10.1111/coa.12878. Epub 2017 Apr 17. PMID 28339165
- [Background] Whitcroft KL, Gunder N, Cuevas M, Andrews P, Menzel S, Haehner A, Hummel T. Intranasal sodium citrate in quantitative and qualitative olfactory dysfunction: results from a prospective, controlled trial of prolonged use in 60 patients. Eur Arch Otorhinolaryngol. 2021 Aug;278(8):2891-2897. doi: 10.1007/s00405-020-06567-7. Epub 2021 Jan 20. PMID 33471169